CLINICAL TRIAL: NCT02192138
Title: Ventilation, Gas Exchange and Cardiac Function in Relation to Intrapleural Pressure Changes in Patients Undergoing Therapeutic Thoracentesis
Brief Title: Pathophysiological Effects of Intrapleural Pressure Changes During Therapeutic Thoracentesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Collaborators: Nalecz Institute of Biocybernetics and Biomedical Engineering, Polish Academy of Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IPU-DIMPA-WUM14(1)
Record Dates: First submitted 2014-07-01; First posted 2014-07-16 (Estimated); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Pleural Effusion; Exudative Pleuritis
Keywords: Pleural effusion; Pleural fluid; Thoracentesis; Intrapleural pressure; Pleural manometry
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Therapeutic thoracentesis (Experimental): Patients with pleural effusion who require therapeutic thoracentesis will be enrolled into the study
  Interventions: Procedure: Therapeutic thoracentesis; Device: Pleural catheter; Device: Pleural manometer

INTERVENTIONS:
Procedure: Therapeutic thoracentesis — Therapeutic thoracentesis with pleural fluid withdrawal
Device: Pleural catheter
Device: Pleural manometer

SUMMARY:
Research project objectives.

The project includes eight research hypotheses and eight corresponding study objectives. The most relevant objectives are:

* Analysis of lung function and gas exchange parameters in relation to the removed pleural fluid volume and intrapleural pressure changes.
* Evaluation of changes in lung and chest wall compliance and related changes in work of breathing during therapeutic thoracentesis and pleural fluid withdrawal.
* Study of the relationship between intrapleural pressure changes and cardiac function assessed by echocardiography and alterations in serum natriuretic peptide A and B concentration.
* Comparative analysis of the reliability of the volume-pressure curve slope prediction based on different variables measured before thoracentesis and real measurements of ventilation and intrapleural pressure during thoracentesis.

  2. Research methodology The study will be performed in 60 patients with pleural effusion planned for therapeutic thoracentesis.

Studies before thoracentesis: body plethysmography, spirometry, lung diffusion capacity (DLCO), arterial blood gases, 6 minute walk test, echocardiography, serum natriuretic peptide concentration.

Evaluation during thoracentesis: continuous measurement of tidal breathing and respiratory rate, measurement of removed pleural fluid volume and intrapleural pressure, transcutaneous measurement of PO2 and PCO2. Pleural catheter will be retained for the next 48hours to enable fluid drainage and intrapleural pressure measurement after completion of thoracentesis.

Monitoring during 48-hrs after thoracentesis: pre-thoracentesis measurements will be repeated in specific time points and compared in two subgroups (active physiotherapy to improve lung re-expansion and passive lung re-expansion).

Intrapleural pressure will be measured 24 and 48 hours after thoracentesis. Then, the catheter will be removed.

Analysis.Signal analysis and visual multidimensional analysis performed with the use of own computer programs will be the first step of the analysis. The identified relationships between the analyzed parameters should allow to form physiological, medical, and statistical hypotheses, as well to verify the analysis of previously obtained data .

Expected impact of the research project The study results will allow to define lung function, blood gases and cardiovascular function in relation to changes in intrapleural pressure. Some of these correlations had not been previously investigated. Our results may influence management standards in patients who require therapeutic thoracentesis.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 - 85 years,
2. pleural effusion occupying more than one third of the hemithorax on the posteroanterior chest radiograph,
3. therapeutic thoracentesis planned on the basis of signs and symptoms as well as imaging and functional studies,
4. no contraindications for thoracentesis,
5. signed informed consent for participation in the study.

Exclusion Criteria:

1. poor performance status requiring maximal shortening of the procedure,
2. instable hemodynamic or respiratory status unrelated to pleural effusion,
3. respiratory failure requiring mechanical ventilation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Change in intrapleural pressure | Continuous measurement as a function of withdrawn pleural fluid during therapeutic thoracentesis - up to 60 minutes
  1) baseline measurement before pleural fluid withdrawal, 2) continuous measurement during pleural fluid withdrawal, 3) measurement 1 minute after termination of pleural fluid withdrawal (the end of the procedure),
Intrapleural pressure | 6 hrs after completion of therapeutic thoracentesis
  Pleural manometer was connected to intrapleural catheter for intrapleural pressure measurement after therapeutic thoracetnesis.

SECONDARY OUTCOMES:
Volume of withdrawn pleural fluid | Continuous measurement during therapeutic thoracentesis - up to 60 minutes
  Continuous measurement during pleural fluid withdrawal, up to the end of the procedure, i.e. approximately 60 minutes

OTHER OUTCOMES:
Change in arterial blood gases and transcutaneous carbon dioxide tension (tcPCO2) and transcutaneous oxygen tension (tcPO2) measurements | Continuous measurement during therapeutic thoracentesis - up to 60 minutes
  1) baseline measurement 5 minutes before pleural fluid withdrawal, 2) continuous measurement during pleural fluid withdrawal, 3) measurement 1 minute after termination of pleural fluid withdrawal (the end of the procedure),
Respiratory pattern including respiratory rate and tidal volume | Continuous measurement during therapeutic thoracentesis - up to 60 minutes
  1) baseline measurement 5 minutes before pleural fluid withdrawal, 2) continuous measurement during pleural fluid withdrawal, 3) measurement 1 minute after termination of pleural fluid withdrawal (the end of the procedure),
Change in lung function | Baseline (approximately 1 hour before thoracentesis) and 6 hrs after therapeutic thoracentesis
  Lung function parameters measured by spirometry and body plethysmography
Change in atrial natriuretic peptide (ANP) and brain natriuretic peptide (BNP) | Baseline (approximately 15 minutes before thoracentesis) and at the end of therapeutic thoracentesis (10 minutes after completion of the procedure, i.e approximately 85 minutes after baseline measurement)
  Venous blood samples were collected for natriuretic peptides measurements.
Arterial blood gases and transcutaneous carbon dioxide tension (tcPCO2) and transcutaneous oxygen tension (tcPO2) measurements | 6 hrs after the completion of therapeutic thoracentesis
  Transcutaneous PO2 and PCO2 were measured in accordance with the manual supplied by the manufacturer of the transcutaneous O2/CO2 monitoring system.
Atrial natriuretic peptide (ANP) and brain natriuretic peptide (BNP) | 6 hrs after the completion of the therapeutic thoracentesis
  Venous blood samples were collected for natriuretic peptides measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Rafal M Krenke, MD, PhD, Principal Investigator — Medical University of Warsaw
Locations (1):
- Medical University of Warsaw, Warsaw, Poland

REFERENCES:
- [Derived] Zielinska-Krawczyk M, Grabczak EM, Michnikowski M, Zielinski K, Korczynski P, Stecka A, Golczewski T, Krenke R. Patterns of pleural pressure amplitude and respiratory rate changes during therapeutic thoracentesis. BMC Pulm Med. 2018 Feb 14;18(1):36. doi: 10.1186/s12890-018-0595-7. PMID 29444649
- [Derived] Zielinska-Krawczyk M, Michnikowski M, Grabczak EM, Palko KJ, Korczynski P, Golczewski T, Krenke R. Cough during therapeutic thoracentesis: friend or foe? Respirology. 2015 Jan;20(1):166-8. doi: 10.1111/resp.12426. Epub 2014 Nov 3. PMID 25367064